CLINICAL TRIAL: NCT00130325
Title: A Double Blind Placebo-controlled Randomized Trial of Isoniazid for the Reversion of a Positive IFNg ELISPOT in TB Case Contacts
Brief Title: A Trial of Isoniazid for the Reversion of Interferon Gamma ELISPOT in Tuberculosis (TB) Case Contacts
Acronym: IRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Research Council Unit, The Gambia (Other)
Responsible Party: Prof. Tumani Corrah, Unit Director, MRC (UK) Laboratories, The Gambia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRS SCC965
Record Dates: First submitted 2005-08-11; First posted 2005-08-15 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Tuberculosis
Keywords: ELISPOT,; tuberculosis,; Mycobacterium tuberculosis; Isoniazid; Clinical trial
MeSH Terms: conditions — Tuberculosis | interventions — Isoniazid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Isoniazid arm
  Interventions: Drug: Isoniazid
- B (Placebo Comparator): Placebo of Isoniazid tablet 300mg
  Interventions: Drug: Placebo of Isoniazid tablets 300mg

INTERVENTIONS:
Drug: Isoniazid — Isoniazid 900mg, tablets, twice a week for 6 months
  Arms: A
Drug: Isoniazid — INH 900mg twice weekly for 6 months
  Arms: A
Drug: Placebo of Isoniazid tablets 300mg — Isoniazid BP 0mg twice weekly for 6 months
  Arms: B

SUMMARY:
There are new TB vaccines already developed that need to be tried in humans to assess their efficacy.

The researchers had previously shown that production of interferon gamma by T cells in response to TB antigens is a more specific marker of TB infection.

The researchers hypothesize that this can be used as a reliable early marker of TB vaccine efficacy. The researchers expect to show a significantly increased reversion of this test in household contacts of TB patients given Isoniazid prophylaxis treatment for 6 months.

DETAILED DESCRIPTION:
Current efforts to control the spread of tuberculosis are failing. An increasingly large number of new generation vaccines are being produced and a plan for assessing their ability to prevent disease and treat infection needs to be developed.

The MRC Labs in The Gambia is well positioned to conduct safety and immunogenicity studies and also to conduct trials of the therapeutic effect of these vaccines in preventing disease in case contacts who are infected.

This study is part one of a three-step plan to develop a reliable early surrogate marker of the therapeutic efficacy of new TB vaccines.

The three-step plan is as follows:

* Evaluate the ability of isoniazid, known to be effective in the treatment of MTB infection, to revert the antigen-specific IFNg-ELISPOT in ESAT-6 and/or CFP-10 positive contacts of TB patients.
* Compare the ability of different combinations of a TB vaccine and isoniazid to revert the ELISPOT in a 4-arm randomised trial using:1) isoniazid alone, 2) a TB vaccine alone, 3) a combination of isoniazid and TB vaccine, and 4) placebo
* Compare, in a randomized trial, the ability of TB vaccine or vaccine plus isoniazid versus isoniazid alone to prevent the development of secondary disease.

For this first step the researchers will test the following hypothesis:

* Those receiving isoniazid have a significantly higher reversion rate of MTB-specific responses as measured with IFNg-ELISPOT assays compared to those who receive a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy person aged 15 years and above
* Normal medical history and physical examination
* Normal biochemistry and haematological indices
* Mantoux ≥ 10mm
* Negative HIV antibody test
* No serological evidence of hepatitis B virus (HBV) infection
* Normal Chest X-ray
* ESAT6 and/or CFP-10 peptides and ESAT6/CFP-10 protein positive (≥10 SFC for ESAT 6 or CFP-10 and ESAT6/CFP-10 protein).
* Index case is sputum smear positive
* Index case has chest X ray (CXR) characteristics of TB

Exclusion Criteria:

* Pregnant female
* Haemoglobin <8 g/dl
* Previous history of tuberculosis
* Clinical case of tuberculosis
* Current participation in another clinical trial, or within 12 weeks of this study.
* Any other factor that might increase the risk of an adverse outcome from participation in the trial
* Significant history or evidence of skin disorder, allergy, immunodeficiency, organ specific disorders causing significant immunodeficiency.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2004-10; Primary Completion 2008-10 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Qualitative IFN-g ELISPOT reversion | 12 months
Quantitative IFN-g ELISPOT reversion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Philip C Hill, MPH FRACP, Principal Investigator — MRC Laboratories, Gambia; Roger H Brookes, PhD, Principal Investigator — MRC laboratories, Gambia; Richard A Adegbola, PhD FRCPath, Study Chair — MRC laboratories, Gambia
Locations (1):
- MRC Laboratories, Banjul, KSMD, The Gambia

REFERENCES:
- [Background] Hill PC, Brookes RH, Fox A, Fielding K, Jeffries DJ, Jackson-Sillah D, Lugos MD, Owiafe PK, Donkor SA, Hammond AS, Otu JK, Corrah T, Adegbola RA, McAdam KP. Large-scale evaluation of enzyme-linked immunospot assay and skin test for diagnosis of Mycobacterium tuberculosis infection against a gradient of exposure in The Gambia. Clin Infect Dis. 2004 Apr 1;38(7):966-73. doi: 10.1086/382362. Epub 2004 Mar 16. PMID 15034828
- [Derived] Adetifa IM, Ota MO, Jeffries DJ, Lugos MD, Hammond AS, Battersby NJ, Owiafe PK, Donkor SD, Antonio M, Ibanga HB, Brookes RH, Aka P, Walton R, Adegbola RA, Hill PC. Interferon-gamma ELISPOT as a biomarker of treatment efficacy in latent tuberculosis infection: a clinical trial. Am J Respir Crit Care Med. 2013 Feb 15;187(4):439-45. doi: 10.1164/rccm.201208-1352OC. Epub 2012 Dec 6. PMID 23220919
- See also: MRC laboratories, Gambia website — http://www.mrc.gm